CLINICAL TRIAL: NCT02280499
Title: Multicenter Clinical Observation PROMOS®
Status: Completed | Type: Observational
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: D8240-1
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-02

CONDITIONS: Primary and Secondary Omarthrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: standard PROMOS prosthesis

SUMMARY:
Overall study design:

This study is a prospective, multicenter, postmarket clinical observation to validate the PROMOS™ Standard Shoulder System as state-of-the-art implant system for total shoulder arthroplasty in terms of radiographic and clinical performance as well as long-term survivorship over 10 years.

DETAILED DESCRIPTION:
Primary objective:

Radiological and clinical loosening rates of the glenoid and humeral components must be comparable or below the rates of other well documented state-of-the-art shoulder systems with cemented glenoid components. Complications occurring intra- or postoperatively will be assessed and sub-classified in their relation to the implant.

At the end of the observation, a long-term survival rate will be calculated according to Kaplan-Meier with revision due to aseptic loosening as the end-point.

Secondary objectives:

The Constant Murley score and the ASES clinical evaluation are used for documenting the improvement in pain, function and range of motion. For the patient's subjective view of improvement in function a patient self-assessment form is used.

ELIGIBILITY:
Inclusion Criteria:

* patient has no general medical contraindication to surgery
* informed consent to participate in the observation signed by the patient
* routine radiographic assessment is possible
* patient is likely to comply with study follow-up requirements
* primary total- or hemi-shoulder-arthroplasty to the affected side, unilateral or bilateral

Exclusion Criteria:

* acute shoulder trauma
* tumor / malignoma
* avascular necrosis
* late stage rotator cuff disease
* Charcot joint disease or other severe neurosensory deficits
* high comorbidity
* previously failed shoulder arthroplasty
* fracture sequelae of proximal humerus
* hypersensitivity to the implant materials used
* addictive disorders such as alcohol or drug abuse
* severe spinal disorders
* bacterial infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2003-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 93 patients were assessed for eligibility. Two participants were excluded before receiving the intervention due to not meeting the inclusion criteria.
  Four enrolled subjects did not receive a PROMOS™ prosthesis due to different reasons but were changed to another shoulder implant which was not part of the study.
Groups:
- Promos™ Standard Shoulder System: All participating subjects underwent primary total shoulder arthroplasty after signing informed consent. All subjects received the Promos™ Standard shoulder system.
Period: Overall Study
Arm/Group | Promos™ Standard Shoulder System
Started | 87
Completed | 26
Not Completed | 61
Not completed — Death | 14
Not completed — Lost to Follow-up | 42
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Arm/Group | Promos™ Standard Shoulder System
Number analyzed (Participants) | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 29
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 26.81 (4.45)

OUTCOME MEASURES:

1. Primary Outcome: Radiological and Clinical Loosening Rates of the Glenoid and Humeral Components
Description: The long-term survival rate of the Promos™ Standard shoulder system was calculated with revision due to aseptic loosening as endpoint using a Kaplan-Meier Analysis.
Time Frame: up to 10 years
Measure: Number (95% Confidence Interval); unit: Percentage survivorship
Arm/Group | Promos™ Standard Shoulder System
Number analyzed (Participants) | 87
Percentage survivorship | 96.29 [85.43 to 99.1]

2. Secondary Outcome: Constant Murley Score
Description: The Constant Murley Score is a shoulder outcome score to determine the functionality of the shoulder after the treatment of a shoulder injury. The score ranges from 0 to 100 with a higher score indicating better shoulder function.
Time Frame: 10 Years
Population: As per the study flow chart, 26 study participants had a 10 year follow-up visit to collect the data supporting the primary outcome measure. The Constant Murley Score was incomplete for 3 participants and therefore the number of participants analyzed is 23.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Promos™ Standard Shoulder System
Number analyzed (Participants) | 23
units on a scale | 72.80 (16.89)

3. Secondary Outcome: ASES Shoulder Score Index
Description: The American Shoulder and Elbow Surgeon's (ASES) evaluation is used to document the improvement in pain, function and range of motion after shoulder injury. The ASES Shoulder Score Index is calculated from the ASES patient related questionnaire and ranges from 0-100 with a higher score indicating improvement in pain and function.
Time Frame: 10Years
Population: As per the study flow chart, 26 study participants had a 10 year follow-up visit to collect the data supporting the primary outcome measure. The ASES Shoulder Score Index was calculated for 27 participants. As the score is a patient reported outcome the score could be completed at home increasing the number of available scores.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Promos™ Standard Shoulder System
Number analyzed (Participants) | 27
units on a scale | 76.88 (18.21)

ADVERSE EVENTS:
Arm/Group | Promos™ Standard Shoulder System
Serious Adverse Events (participants affected / at risk) | 31/87
Other Adverse Events (participants affected / at risk) | 2/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Promos™ Standard Shoulder System (N=87)
Partial Plexus paresis (Nervous system disorders) | 1
Fall - traum. rupture of subscapularis (Musculoskeletal and connective tissue disorders) | 1
Total shoulder arthroplasty contralateral side (Musculoskeletal and connective tissue disorders) | 1
Stroke (Blood and lymphatic system disorders) | 1
Pulmonary Embolism (Blood and lymphatic system disorders) | 1
Heart attack (Blood and lymphatic system disorders) | 2
Trauma (abduction and rotation) (Musculoskeletal and connective tissue disorders) | 1
Pneumonia (Infections and infestations) | 1
Migration of humeral component (Musculoskeletal and connective tissue disorders) | 1 — Rotator cuff led to sup. migration of humeral component
Thrombosis right leg (Blood and lymphatic system disorders) | 1
Glenoid loosening (Musculoskeletal and connective tissue disorders) | 1
Death (General disorders) | 14
Revision of study device (Investigations) | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Promos™ Standard Shoulder System (N=87)
Subacromial Impingement (Musculoskeletal and connective tissue disorders) | 1
No active mobilization after surgery due to pain (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
One limitation of the study relates to the small number of subjects available at the 10 year interval for final analysis due to the early termination of 2 sites.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No